CLINICAL TRIAL: NCT04060576
Title: Post-Needling Soreness Depending On The Needle Diameter On Dry Needling On The Most Hyperalgesic Area Of The Internal Gastrocnemius In Plantar Fasciitis: A Randomised Controlled Trial
Brief Title: Post-needling Soreness After Internal Gastrocnemius Muscle Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Dr. Daniel Pecos Martín, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIM/HU/2019/01
Record Dates: First submitted 2019-08-14; First posted 2019-08-19 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Heel Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A treated with a 16-gauge needle (Experimental): Group A is intervened on the gastrocnemius muscle with a 16-gauge needle.
  Interventions: Procedure: Dry needling treatment with a thinner needle
- Group B treated with a 25-gauge needle (Experimental): Group B is intervened on the gastrocnemius muscle with a 25-gauge needle.
  Interventions: Procedure: Dry needling treatment with a medium-sized needle
- Group C treated with a 32-gauge needle (Experimental): Group C is intervened on the gastrocnemius muscle with a 32-gauge needle.
  Interventions: Procedure: Dry needling treatment with a thickest needle

INTERVENTIONS:
Procedure: Dry needling treatment with a thinner needle — We will make an application with the dry needling technique with a fine needle on the myofascial trigger points of the gastrocnemius muscle.
  Arms: Group A treated with a 16-gauge needle
Procedure: Dry needling treatment with a medium-sized needle — We will make an application with the dry needling technique with a medium-sized needle on the myofascial trigger points of the gastrocnemius muscle.
  Arms: Group B treated with a 25-gauge needle
Procedure: Dry needling treatment with a thickest needle — We will make an application with the dry needling technique with the thickest needle on the myofascial trigger points of the gastrocnemius muscle.
  Arms: Group C treated with a 32-gauge needle

SUMMARY:
Mechanical hyperalgesia areas, also known as myofascial trigger points, are treated by manual therapy or invasive technics. Dry needling achieves an improvement of the symptomatology in 70% of the subjects, being the acute patients the most benefited. However, bruising, bleeding, pain during treatment or post-needling soreness. Plantar fasciitis is the most common cause of interior heel pain, affects approximately 10% of the general population and is one of the most benefited pathologies in the long term by the application of dry needling The gauge of the needle chosen for the treatment can influence post-needling soreness intensity and pressure pain threshold.

Objective To evaluate the relation between post-needling soreness intensity and needle diameter on the treatment of the most hyperalgesic point of the internal gastrocnemius.

Hypothesis Post-needling soreness intensity and pressure pain threshold depend on needle diameter applied in the treatment of the most hyperalgesic point of the internal gastrocnemius.

DETAILED DESCRIPTION:
Intervention:

Two zones are established:

* Zone 1: where researcher nº 1 controls the data management and sample randomization.
* Zone 2: where researcher nº 2 locates the most hyperalgesic area and measures pressure point threshold variable and researcher nº 3 performs dry needling puncture.

Researcher nº 1 explains to the subjects how the study works, collects the confidential documents and scores the independent variables (sex, age and BMI). Every subject receives an identification code and is randomly assign to a intervention group (A, B or C) Researcher nº 2 makes delivery of the document where the variables pressure pain threshold and post-needling soreness intensity will be written down. Firstly, the visual analogue scale compliance prior to the intervention is requested. After that, the subject is placed in prone position on the stretcher with a slight knee flexion and the most hyperalgesic area in the internal gastrocnemius of the lower limb with plantar fasciitis is located and marked.

Researcher nº 2 performs the algometry at the most hyperalgesic area (3 measurements with 30 seconds between them), writes down the results of pressure pain threshold variable and leaves the room.

Researcher nº 3 receives a needle from researcher nº 1 ignoring its diameter (colour tab is removed). Firstly, contamination is prevented by disinfection, then, 10 insertions are made at the marked point (the number of local twitch response are counted) and the needle used is thrown in the sanitary waste container. Ischemic compression is performed for 60 seconds followed by an analytical stretch of the internal gastrocnemius for 30 seconds.

Once researcher nº 3 has finished the intervention leaves the room and researcher nº 2 returns to repeat the measurements (post-needling soreness intensity, by filling in VAS, and pressure pain threshold, performing algometry).

Researcher nº 2 reminds the subject to complete VAS at 12, 24, 48 and 72 hours (suggesting setting an alarm) and makes an appointment 48 hours after to perform the third measure of pressure pain threshold variable.

When all the data needed for the study has been collected, researcher nº1 gathers results and exports them for statistical interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65.
* Plantar Fasciitis diagnosis.
* Presence of hyperalgesic area in the internal gastrocnemius.

Exclusion Criteria:

* Belenophobia
* Hypothyroidism Presence of hyperalgesic area in the internal gastrocnemius - Diabetes
* Lymphedema o lymphatic surgery Muscle diseases
* Anticoagulant consumption Knee or ankle surgery
* Analgesic consumption during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Post-needling soreness intensity | Change From Baseline in Pain Scores on the Visual Analog Scale at 72 hours.
  The investigators use a Visual Analog Scale (VAS) to determine the intensity of the patient's post-needing pain after and for 72 hours after DN.The VAS is a 100-mm line, oriented horizontally, with one end representing "no pain" and the other end representing "worst pain." Subjects will be asked to rate their current pain with a mark on the scale.
Pressure Pain Threshold | Change from Baseline Pressure Pain Threshold at 72 hours
  The PPT serves to determine the sensitivity of hiperalgesic focus. The investigators will done it with one algometer. A lower threshold is a worse result. A higher threshold is a better result.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Gallego-Izquierdo, Dr, Study Chair — Alcala University
Locations (2):
- Spain (2):
  - Instituto Fisioterapia y Dolor, Alcalá de Henares, Madrid
  - Grupo Fisioterapia y Dolor, Alcalá de Henares, Madrid